CLINICAL TRIAL: NCT03222037
Title: Evaluation of Electronic LogMar Visual Acuity and Contrast Sensitivity in a Population of Contact Lens Wearers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5968
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2018-08-24 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/SCR (Experimental): Subjects who are current soft contact lens wearers between the ages of 18 and 35 will be randomized to the two different treatments (TEST/SCR) sequentially
  Interventions: Device: senofilcon A; Device: Control
- SCR/TEST (Experimental): Subjects who are current soft contact lens wearers between the ages of 18 and 35 will be randomized to the two different treatments (SCR/TEST) sequentially
  Interventions: Device: senofilcon A; Device: Control

INTERVENTIONS:
Device: senofilcon A — Acuvue Oasys 1-Day
Device: Control — Trial Frame with best spherocylindrical refraction (SCR)

SUMMARY:
This is a bilateral, non-dispensing, randomized, cross-over, single-masked study. There are a total of 3 visits where all study endpoints will be measured in all subjects at baseline with habitual lenses and under the two testing treatments sequentially in separate visits based on the randomization scheme

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol
3. Between 18 and 35 (inclusive) years of age at the time of screening
4. The subject must be habitual contact lens wearers (defined as minimum 6 hours per day, 5 days a week over the last month)
5. The subject must meet all of the following three criteria:

   1. The eyes' spherical equivalent distance refraction must be in the range of -1.00 to -9.00 D (inclusive)
   2. The eyes' refractive cylinder must be less than or equal to -0.75 DC
   3. Each eye must have best corrected visual acuity of 20/25 or better.
6. The subject must have normal eyes (i.e., no ocular medications or infections of any type)

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Currently pregnant or lactating
2. Any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study
3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear or may impact the functioning of the tear film (e.g., Isotretinoin)
4. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion
5. Any current use of ocular medication
6. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
7. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the Efron scale
8. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear
9. Any known hypersensitivity or allergic reaction to contact lens care products.
10. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment
11. Employee of clinical site (e.g., Investigator, Coordinator, Technician)
12. Current wearers of Acuvue Oasys 1-Day brand contact lenses

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VRC East, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 49 subjects were enrolled into this study. Of the enrolled subjects, 43 were dispensed at least one study article. Of the dispensed subjects all 43 completed the study.
Groups:
- Test/SCR: Subjects that were randomized to receive the Test lens during the first period and then the SCR (Subjective Spherorcylindrical Refraction) treatment during the second period.
- SCR/Test: Subjects that were randomized to receive the SCR (Subjective Spherorcylindrical Refraction) treatment during the first period and then the Test lens during the second period.
Period: Period 1
Arm/Group | Test/SCR | SCR/Test
Started | 21 | 22
Completed | 21 | 22
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test/SCR | SCR/Test
Started | 21 | 22
Completed | 21 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Dispensed: All subjects dispensed at least one study treatment.
Arm/Group | Total Dispensed
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.8 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 7
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Asian | 8
  Black or African American | 6
  White | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (logMAR)
Description: Visual Acuity was collected electronically under two conditions (high luminance low contrast and low luminance high contrast) in both eyes 15- minutes post study article administration. The average visual acuity for each lens type and condition was reported.
Time Frame: 15 Minutes post Treatment Administration
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Test: Subjects that received the Test lens during either the first or second period of the study.
- SCR (Subjective Spherorcylindrical Refraction): Subjects that received the SCR treatment during either the first or second period of the study.
Arm/Group | Test | SCR (Subjective Spherorcylindrical Refraction)
Number analyzed (Participants) | 43 | 43
Number analyzed (Eyes) | 86 | 86
logMAR
  High Luminance Low Contrast | 0.15 (0.108) | 0.21 (0.130)
  Low Luminance high Contrast | 0.02 (0.097) | 0.05 (0.102)
Statistical Analysis 1: Comparison: Test vs SCR (Subjective Spherorcylindrical Refraction); Comparison between the Test and the SCR treatments was carried out using 97.5% confidence intervals for the least-square mean differences; Test type: Non-Inferiority — Non-inferiority was declared if the upper limit of the 97.5% confidence interval was below 0.05; Linear Mixed Model; Linear mixed model with Kenward and Roger method for degrees of freedom; Mean Difference (Final Values) = -0.06, 97.5% CI 2-sided [-0.09 to -0.02], Standard Error of Mean 0.02 — Mean difference was calculated as Test- SCR. This comparison is for high lumniance low contrast
Statistical Analysis 2: Comparison: Test vs SCR (Subjective Spherorcylindrical Refraction); Test type: Non-Inferiority — Non-inferiority was declared if the upper limit of the 97.5% confidence interval was below 0.05; Linear Mixed Model; Linear mixed model with Kenward and Roger method for denominator degrees of freedom; Median Difference (Final Values) = -0.03, 97.5% CI 2-sided [-0.06 to -0.01], Standard Error of Mean 0.01 — Mean difference was calculated as Test- SCR. This comparison is for Low luminance high contrast

2. Secondary Outcome: Area Under Contrast Sensitivity Function Curve
Description: Contrast sensitivity was assessed in both eyes at 1.5, 3.0, 6.0, 12.5 and 18.0 cycles per degrees (cpd) using AST Sentio vision Testing System. During testing 25 triplets of test letters were displayed on a large stationary monitor (118 CM), the operator recorded the patients responses using the remote (Android Tablet). After a testing session had been completed the software calculated the Area under the log contrast sensitivity function from 1.5 cpd to 18 cpd.
Time Frame: 15 minutes post treatment administration
Population: All subjects who completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: log
Units Other Than Participants: Eyes
Arm/Group | Test | SCR (Subjective Spherorcylindrical Refraction)
Number analyzed (Participants) | 43 | 43
Number analyzed (Eyes) | 86 | 86
log | 1.39 (0.135) | 1.34 (0.185)
Statistical Analysis 1: Comparison: Test vs SCR (Subjective Spherorcylindrical Refraction); Comparison between the Test and SCR treatments was carried out using least-square mean differences; Test type: Equivalence — Statistical significance is declared if the lower limit of the 95% confidence interval is above 0 or if the upper limit of the 95% confidence interval is below 0; p = 0.0066, Linear Mixed Model; Linear Mixed Model with Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0.01 to 0.08], Standard Error of Mean 0.02 — Mean difference was calculated as Test - SCR

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 2 weeks per subject.
Arm/Group | Test | SCR (Subjective Spherorcylindrical Refraction)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT03222037/Prot_SAP_000.pdf